CLINICAL TRIAL: NCT06409481
Title: Pharmacovigilance Assessment of Reporting of Cardiovascular Adverse Events With Antineoplastic Agents (PARCA)
Acronym: PARCA
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: EC-024-092
Record Dates: First submitted 2024-04-25; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Cardiac Diseases; Vascular Diseases; Cancer
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Vascular Diseases; Neoplasms | interventions — Antineoplastic Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Adverse Events with Antineoplastic agents: Cases reported in VigiBase, FAERS and other pharmacovigilance databases of patients treated by antineoplastic agents, with a chronology compatible with the drug toxicity.
  Interventions: Drug: Antineoplastic Agents

INTERVENTIONS:
Drug: Antineoplastic Agents — small-molecule kinase inhibitors, immune checkpoint inhibitors, monoclonal antibodies, cytotoxic drugs, and other therapeutics

SUMMARY:
The aim of this observational study is to explore and analyze reports of cardiac or vascular adverse events linked to the administration of antineoplastic agents among patients diagnosed with tumors represented by advanced non-small cell lung cancer. The study leverages pharmacovigilance databases such as the World Health Organization (WHO) database (VigiBase), FDA Adverse Event Reporting System (FAERS), and others to gather individual safety case reports for analysis.

DETAILED DESCRIPTION:
Concomitant antineoplastic drug therapy may produce serious adverse cardiac or vascular system events. In this study, reports of cardiovascular adverse drug events following treatment with antineoplastic drugs were investigated using the World Health Organization (WHO) personal safety case report database (VigiBase) and FDA Adverse Event Reporting System (FAERS).

ELIGIBILITY:
Inclusion Criteria:

1. Case reported in VigiBase, FAERS and other pharmacovigilance databases of individual safety case reports to 12/31/2024.
2. Adverse events reported were including the MedDRA terms: Cardiac disorders (SOC), Vascular disorders (SOC), Cardiac and vascular investigations (excl enzyme tests) (HLGT), Sudden death (PT), Sudden cardiac death (PT), Cardiac arrhythmias (HLGT), Cardiac disorder signs and symptoms (HLGT), Cardiac neoplasms (HLGT), Cardiac valve disorders (HLGT), Coronary artery disorders (HLGT), Endocardial disorders (HLGT), Heart failures (HLGT), Myocardial disorders (HLGT), Pericardial disorders (HLGT), Vascular disorders NEC(HLGT), Vascular inflammations(HLGT), Embolism and thrombosis(HLGT), Vascular hypertensive disorders(HLGT), Blood pressure disorders NEC(HLGT), Venous varices(HLGT), Arteriosclerosis, stenosis, vascular insufficiency and necrosis(HLGT), Aneurysms and artery dissections(HLGT).
3. Patients treated with antineoplastic agents (including small-molecule kinase inhibitors, immune checkpoint inhibitors, monoclonal antibodies, cytotoxic drugs, and other therapeutics).
4. The number of reports corresponding to each drug or adverse event is at least three.
5. The primary indication is malignant tumors, specifically advanced non-small cell lung cancer.

Exclusion Criteria:

1. Any of the information in the baseline information such as gender, age, region, date of report is empty.
2. The severity level of the reported adverse event is empty.
3. Adverse events were reported in patients whose drug indications included cardiovascular disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been treated with an antineoplastic agent and have been diagnosed with tumors that represent advanced non-small cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 800000 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Cardio-vascular toxicity of antineoplastic agents | Case reported in VigiBase, FAERS and other pharmacovigilance databases of individual safety case reports to 12/31/2024
  Identification and report of the cardio-vascular toxicity of antineoplastic agents. The research includes the report with MedDRA terms: SOC Cardiac Disorders, SOC Vascular Disorders, Cardiac and vascular investigations (excl enzyme tests) (HLGT), Skeletal and cardiac muscle analyses (HLT), Sudden death (PT). Drugs investigated are antineoplastic agents.

SECONDARY OUTCOMES:
Causality assessment of reported cardiovascular events according to pharmacovigilance databases | Case reported in VigiBase, FAERS and other pharmacovigilance databases of individual safety case reports to 12/31/2024
  Disproportionality individual case data analysis between cardiovascular events and antineoplastic agents.
Assessment of the association between cardiovascular toxicity due to antineoplastic agents and risk factors. | Case reported in VigiBase, FAERS and other pharmacovigilance databases of individual safety case reports to 12/31/2024
  Cardiovascular events are identified using MedDRA terms. Each cardiovascular event and risk factor will be assessed for potential over-reporting by calculating odds ratios. Factors evaluated will include, but are not limited to, cancer type and patient baseline characteristics (gender, age, country of reporting, etc.). Additionally, the year of reporting and other relevant variables will be considered.
Assess cardiovascular toxicity differences among antineoplastic agent classes and within the same class. | Case reported in VigiBase, FAERS and other pharmacovigilance databases of individual safety case reports to 12/31/2024
  The data were classified into different drug classes based on the Anatomical Therapeutic Chemical (ATC) classification system. This included small molecule kinase inhibitors, immune checkpoint inhibitors, and monoclonal antibodies. The occurrence of major adverse events was identified using the Medical Dictionary for Regulatory Activities (MedDRA) terminology. The differences in cardiovascular toxicity between drug classes were evaluated using disproportionality analysis (single drug vs. full database). To assess toxicity differences between drugs in the same class, for example, a comparison could be made between the cardiovascular toxicity of drugs such as erlotinib, afatinib, and osimertinib, which all belong to the category of EGFR tyrosine kinase inhibitors. Disproportionality analyses (single drug vs. other drugs in the same class) were employed in this regard.
Assessment of the severity of cardiovascular toxicity associated with antineoplastic agents | Case reported in VigiBase, FAERS and other pharmacovigilance databases of individual safety case reports to 12/31/2024
  Reports with fatal outcomes will be compared with reports without fatal outcomes. Odds ratio will be calculated to compare covariates that may be associated with an increased risk of death, including type of adverse cardiovascular event, type of cancer reported, age of the patient, gender, comorbidities, and antitumor monotherapy or combination therapy.
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | Case reported in VigiBase, FAERS and other pharmacovigilance databases of individual safety case reports to 12/31/2024
  The analysis includes analyzing the relationship between the duration of treatment and the occurrence of toxicity, taking into account the cumulative dose of the administered medication.
Description of the drug-drug interactions associated with adverse events. | Case reported in VigiBase, FAERS and other pharmacovigilance databases of individual safety case reports to 12/31/2024
  Describe cardiovascular adverse events reported when two or more drugs are taken concurrently or consecutively in patients with the same indication.
Description of the population of patients having a cardio-vascular adverse events | Case reported in VigiBase, FAERS and other pharmacovigilance databases of individual safety case reports to 12/31/2024
  The patient population with cardiovascular adverse events was described in terms of baseline information, including patient indication, age, sex, country of reporting origin, and clinical outcomes, among other factors.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Kang, PhD, Study Director — First Affiliated Hospital of Xinjiang Medical University

IPD SHARING:
Plan to Share IPD: No